CLINICAL TRIAL: NCT04565756
Title: A Randomised, Double-Masked Vehicle-Controlled, Multiple Dose, Dose Escalation Study To Evaluate The Safety and Tolerability of EXN407 in Subjects With Centre Involved Diabetic Macular Oedema Secondary to Diabetes Mellitus
Brief Title: A Study to Evaluate the Safety and Tolerability of EXN407
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Exonate Limited (Industry)
Collaborators: Novotech (Australia) Pty Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Treatment
Other Study IDs: PQ-110-001
Record Dates: First submitted 2020-08-26; First posted 2020-09-25 (Actual); Results first posted 2025-05-09 (Actual); Last update posted 2025-05-09 (Actual); Status verified 2025-04

CONDITIONS: Diabetic Macular Edema

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Dose Escalation Cohort 1 (Experimental): Each subject will receive a low-dose 0.5 mg/mL (0.05%) of EXN407 or placebo twice a day in 14 doses over a 7 day period.
  Interventions: Drug: EXN407
- Dose Escalation Cohort 2 (Experimental): Each subject will receive a mid-dose 1 mg/mL (0.1%) of EXN407 or placebo twice a day in 14 doses over a 7 day period.
  Interventions: Drug: EXN407
- Dose Escalation Cohort 3 (Experimental): Each subject will receive a high-dose 1.5 mg/mL (0.15%) of EXN407 or placebo twice a day in 14 doses over a 7 day period.
  Interventions: Drug: EXN407
- Dose Expansion Cohort (Experimental): The highest well-tolerated dose of EXN407 will be evaluated where subjects will receive EXN407 at the selected dose or placebo twice a day for up to 84 days resulting in a total of 168 doses
  Interventions: Drug: EXN407

INTERVENTIONS:
Drug: EXN407 — EXN407 or placebo will be administered as a single 30 microliters drop twice a day, by unilateral eye drop administration to the study eye only.

SUMMARY:
This first in human (FIH), Phase Ib/II study of EXN407 is a randomised, double-masked, vehicle-controlled, multiple dose, dose-escalating study to evaluate the safety and tolerability of EXN407 in subjects with centre involved Diabetic Macular Oedema (DMO), with Centre-subfield macular thickness (CMT) between 280-420 µm and Best corrected visual acuity (BCVA) better than or equal to 69 ETDRS score (approximate Snellen equivalent 20/40 (6/12 letters) in the study eye, which is considered secondary to diabetes mellitus.

This study will provide a basis for further clinical development of EXN407 ophthalmic solution.

DETAILED DESCRIPTION:
EXN407 or vehicle-control solution administered unilaterally to the study eye only. To select the study eye the Investigator examines the subjects and identifies which eye exhibits centre involved DMO with a CMT between 280-420 μm (as determined by SD-OCT). Further, all other inclusion/exclusion criteria required to be met.

Dose Escalation Cohorts The study assesses the safety and tolerability of EXN407 in eligible subjects with center involved Diabetic Macular Oedema (DMO) at up to 3 escalating dose (concentration) levels and placebo (vehicle) consisting of an excipient formulation adjusted for osmolality. EXN407 or vehicle-control administered as a single 30 μL drop by unilateral eye drop administration to the study eye only, and the drops dosed BID for 7 days. Subjects assessed throughout the treatment period for safety, tolerability, and efficacy at Follow-up visits. Each of the ascending dose subject cohorts consists of 4 subjects (3 subjects randomised to receive EXN407 and 1 subject randomised to receive placebo).

Dose Expansion Cohort The highest well tolerated dose of EXN407 (as recommended by the DEC) is evaluated in a subject expansion cohort in eligible subjects with center involved Diabetic Macular Oedema (DMO) which consists of up to a maximum of 40 subjects (randomised to receive EXN407 at the selected dose or vehicle at a 2:1 drug: placebo ratio). Each eligible subject in the expansion cohort to receive study drug for up to 84 days, resulting in a total of 168 doses (168 single drops of 30 μL volume) of EXN407 or vehicle.

ELIGIBILITY:
Inclusion Criteria:

1. Subject is at least 18 years of age inclusive, at the time of signing the informed consent.
2. BCVA better than or equal to 69 ETDRS score (approximate Snellen equivalent 20/40 or 6/12) in the study eye using the ETDRS visual acuity scale at Screening or BCVA less than 69 ETDRS score (approximate Snellen equivalent 20/50 or 6/15) but who, in the Investigator's opinion, is unsuitable for treatment with anti-VEGF by intravitreal injection or refuses it. Subjects should have no more than a 7-letter difference in BCVA at Screening and baseline visit.
3. Ocular media is consistent with SD-OCT imaging and cataracts are not expected in the subject for the duration of the study.
4. The subject has no other retinal disease.
5. Subject or the subject's partner successfully demonstrates their ability to self-administer/administer eye drops at Screening, with multiple attempts allowed at the discretion of the Investigator.

Exclusion Criteria:

1. Any other retinal disease in the study eye, other than centre involved DMO or diabetic retinopathy.
2. Poor vision (VA 6/60 or worse) in the contralateral eye.
3. Intraocular inflammation (including trace or greater) in the study eye. History of idiopathic or autoimmune uveitis in either eye.
4. Use of intravitreal anti-VEGF drugs including ranibizumab, bevacizumab, aflibercept in the study eye within 6 months of the Screening Visit, or in the fellow (non study) eye within 3 months of the Screening Visit. Use of topical corticosteroids or topical non-steroidal anti-inflammatory agents in the study eye within 28 days of the Screening Visit. Use of intravitreal corticosteroids in either eye or systemic steroids within 12 months of the Screening Visit. Prior use of Iluvien (without time limitation).
5. Within 180 days prior to the Screening visit, use of medications known to be toxic to the retina, lens or optic nerve (e.g. desferoximine, chloroquine/hydrochloroquine, chlorpromazine, phenothiazines, tamoxifen, and ethambutol).
6. History of (within 90 days of Screening date) cerebral vascular accident (stroke) or MI.
7. Significant renal impairment including subjects on chronic renal dialysis and subjects with a history of nephrectomy or kidney transplant (regardless of renal function).
8. History of anaphylaxis, anaphylactoid (resembling anaphylaxis) reactions, or severe allergic responses.
9. Positive pregnancy test (all female subjects of childbearing potential must have a urine β-human chorionic gonadotropin [hCG] pregnancy test performed at Screening and within 7 days prior to randomisation) or is known to be pregnant or lactating.
10. Known to have, or history of a positive test result for, hepatitis B or C, HIV, syphilis, tuberculosis, or COVID-19.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2020-11-05 (Actual); Primary Completion 2022-10-25 (Actual); Study Completion 2022-11-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mark Gillies, Prof, Principal Investigator — Sydney Eye Hospital/Save Sight Institution; Andrew Chang, A/Prof, Principal Investigator — Sydney Retina Clinic & Day Surgery; Sanjeewa Wickremasinghe,, Prof, Principal Investigator — Centre for Eye Research Australia (CERA); Fred Chen, Dr, Principal Investigator — Lions Eye Institute; Jolly Gilhotra, A/Prof, Principal Investigator — Adelaide Eye and Retina Centre; Wilson Heriot, A/Prof, Principal Investigator — ZAVe Clinical Research Management - Retinology Institute; Hemal Mehta, Dr, Principal Investigator — Strathfield Retina Clinic; Peter Davies, Dr, Principal Investigator — Newcastle Eye Hospital Foundation; Rohan Merani, Dr, Principal Investigator — Macquarie University; Helene Cass, Dr, Principal Investigator — Marsden Eye Specialists; Lily Ooi, Principal Investigator — Princess Alexandra Hospital
Locations (11):
- Australia (11):
  - Macquarie University, Macquarie, New South Wales
  - Marsden Eye Specialists, Parramatta, New South Wales
  - Sydney Eye Hospital/Save Sight Institution, Sydney, New South Wales
  - Strathfield Retina Clinic, Sydney, New South Wales
  - Newcastle Eye Hospital Foundation, Waratah, New South Wales
  - Princess Alexandra Hospital, Woolloongabba, Queensland
  - Adelaide Eye and Retina Centre, Adelaide, South Australia
  - Centre for Eye Research Australia (CERA), Melbourne, Victoria
  - Retinology Institute, Melbourne, Victoria
  - Lions Eye Institute, Nedlands, Western Australia
  - Sydney Retina Clinic & Day Surgery, Sydney

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Dose Escalation EXN407 Cohort 1: Each subject will receive a low-dose 0.5 mg/mL (0.05%) of EXN407 or placebo twice a day in 14 doses over a 7 day period.
  EXN407: EXN407 or placebo will be administered as a single 30 microliters drop twice a day, by unilateral eye drop administration to the study eye only.
- Dose Escalation EXN407 Cohort 2: Each subject will receive a mid-dose 1 mg/mL (0.1%) of EXN407 or placebo twice a day in 14 doses over a 7 day period.
  EXN407: EXN407 or placebo will be administered as a single 30 microliters drop twice a day, by unilateral eye drop administration to the study eye only.
- Dose Escalation EXN407 Cohort 3: Each subject will receive a high-dose 1.5 mg/mL (0.15%) of EXN407 or placebo twice a day in 14 doses over a 7 day period.
  EXN407: EXN407 or placebo will be administered as a single 30 microliters drop twice a day, by unilateral eye drop administration to the study eye only.
- Dose Escalation Pooled Placebo Cohort: Data from the placebo subjects in the 3 dose escalation groups was pooled giving a total of n=4
- Dose Expansion EXN407 Cohort: The highest well-tolerated dose of EXN407 will be evaluated where subjects will receive EXN407 at the selected dose or placebo twice a day for up to 84 days resulting in a total of 168 doses
  EXN407: EXN407 or placebo will be administered as a single 30 microliters drop twice a day, by unilateral eye drop administration to the study eye only.
- Dose Expansion Placebo Cohort: Dose expansion cohort consisted of subjects randomised to receive EXN407 at the selected dose or placebo (vehicle) at a 2:1 drug: placebo ratio.
Period: Overall Study
Arm/Group | Dose Escalation EXN407 Cohort 1 | Dose Escalation EXN407 Cohort 2 | Dose Escalation EXN407 Cohort 3 | Dose Escalation Pooled Placebo Cohort | Dose Expansion EXN407 Cohort | Dose Expansion Placebo Cohort
Started | 3 | 3 | 3 | 4 | 23 | 12
Completed | 3 | 3 | 3 | 4 | 22 | 11
Not Completed | 0 | 0 | 0 | 0 | 1 | 1
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 1 | 0
Not completed — Protocol Violation | 0 | 0 | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Dose Escalation EXN407 Cohort 1 | Dose Escalation EXN407 Cohort 2 | Dose Escalation EXN407 Cohort 3 | Dose Escalation Pooled Placebo Cohort | Dose Expansion EXN407 Cohort | Dose Expansion Placebo Cohort | Total
Number analyzed (Participants) | 3 | 3 | 3 | 4 | 23 | 12 | 48
Age, Continuous [Median (Full Range); unit: years] | 60 [55 to 76] | 60 [57 to 73] | 67 [61 to 75] | 59 [49 to 73] | 63 [40 to 78] | 59 [47 to 81] | 61 [40 to 81]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 1 | 0 | 2 | 7 | 4 | 14
  Male | 3 | 2 | 3 | 2 | 16 | 8 | 34
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 0 | 0 | 0 | 0 | 3 | 3 | 6
  Black or African American | 0 | 0 | 0 | 1 | 0 | 0 | 1
  White | 3 | 2 | 2 | 3 | 18 | 9 | 37
  Other | 0 | 1 | 1 | 0 | 2 | 0 | 4
Region of Enrollment [Number; unit: participants]
  Australia | 3 | 3 | 3 | 4 | 23 | 12 | 48
BCVA [Mean (Standard Deviation); unit: BCVA (Letters)] | 83.3 (3.51) | 83.0 (1.00) | 71.3 (1.53) | 86.3 (5.56) | 81.3 (6.04) | 83.6 (7.44) | 82.1 (6.54)
Corneal thickness [Mean (Standard Deviation); unit: microns] | 561.3 (62.80) | 526.3 (10.02) | 581.7 (53.31) | 565.8 (25.86) | 555.6 (33.75) | 548.5 (38.35) | 553.2 (34.99)

OUTCOME MEASURES:

1. Primary Outcome: The Primary Objective of the Study is to Evaluate the Ocular Safety and Tolerability (by Incidence of Ocular Adverse Events) of EXN407 Ophthalmic Solution in Dose Escalation Phase.
Description: Number of Participants with Ocular Treatment Emergent Adverse Events (TEAEs)
Time Frame: Assessed starting from Day 1 of treatment to Day 36 in Dose Escalation.
Population: The Safety population comprised all randomised subjects who received any amount of study drug. Summaries, listings, and analyses were based on the treatment actually received. Screen failures and randomised subjects who did not receive any medication were excluded from the safety analysis set.
  The Safety population was used for the summaries of all safety assessments.
Measure: Count of Participants; unit: Participants
Groups:
- Dose Escalation EXN407 Cohort 1 Study Eye; Dose Escalation EXN407 Cohort 1 Contralateral Eye; Dose Escalation EXN407 Cohort 1, Bilateral Eye: Each subject will receive a low-dose 0.5 mg/mL (0.05%) of EXN407 or placebo twice a day in 14 doses over a 7 day period.
  EXN407: EXN407 or placebo will be administered as a single 30 microliters drop twice a day, by unilateral eye drop administration to the study eye only.
- Dose Escalation EXN407 Cohort 2 Study Eye; Dose Escalation EXN407 Cohort 2 Contralateral Eye; Dose Escalation EXN407 Cohort 2 Bilateral Eye: Each subject will receive a mid-dose 1 mg/mL (0.1%) of EXN407 or placebo twice a day in 14 doses over a 7 day period.
  EXN407: EXN407 or placebo will be administered as a single 30 microliters drop twice a day, by unilateral eye drop administration to the study eye only.
- Dose Escalation EXN407 Cohort 3 Study Eye; Dose Escalation EXN407 Cohort 3 Contralateral Eye; Dose Escalation EXN407 Cohort 3 Bilateral Eye: Each subject will receive a high-dose 1.5 mg/mL (0.15%) of EXN407 or placebo twice a day in 14 doses over a 7 day period.
  EXN407: EXN407 or placebo will be administered as a single 30 microliters drop twice a day, by unilateral eye drop administration to the study eye only.
- Pooled Placebo (Cohort 1, Cohort 2, Cohort 3) Study Eye; Pooled Placebo (Cohort 1, Cohort 2, Cohort 3) Contralateral Eye; Pooled Placebo (Cohort 1, Cohort 2, Cohort) Bilateral Eye: Data from the placebo subjects was pooled (as appropriate).
Arm/Group | Dose Escalation EXN407 Cohort 1 Study Eye | Dose Escalation EXN407 Cohort 1 Contralateral Eye | Dose Escalation EXN407 Cohort 1, Bilateral Eye | Dose Escalation EXN407 Cohort 2 Study Eye | Dose Escalation EXN407 Cohort 2 Contralateral Eye | Dose Escalation EXN407 Cohort 2 Bilateral Eye | Dose Escalation EXN407 Cohort 3 Study Eye | Dose Escalation EXN407 Cohort 3 Contralateral Eye | Dose Escalation EXN407 Cohort 3 Bilateral Eye | Pooled Placebo (Cohort 1, Cohort 2, Cohort 3) Study Eye | Pooled Placebo (Cohort 1, Cohort 2, Cohort 3) Contralateral Eye | Pooled Placebo (Cohort 1, Cohort 2, Cohort) Bilateral Eye
Number analyzed (Participants) | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 4 | 4 | 4
Participants | 2 | 2 | 2 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Statistical Analysis 1: Comparison: Dose Escalation EXN407 Cohort 1 Study Eye vs Dose Escalation EXN407 Cohort 2 Study Eye vs Dose Escalation EXN407 Cohort 3 Study Eye vs Pooled Placebo (Cohort 1, Cohort 2, Cohort 3) Study Eye; Since the primary objective of the study was to evaluate ocular safety and tolerability, no formal hypothesis testing was performed for any continuous or categorical variables. All statistical analyses were descriptive in nature and any statistical inferences were carried out according to the analysis plan and interpreted in view of the exploratory nature of the study; Test type: Other; Since the primary objective of the study was to evaluate ocular safety and tolerability, no formal hypothesis testing was performed for any continuous or categorical variables

2. Primary Outcome: The Primary Objective of the Study is to Evaluate the Ocular Safety and Tolerability (by Incidence of Ocular Adverse Events) of EXN407 Ophthalmic Solution in Dose Expansion Phase.
Description: Number of Participants with Ocular Treatment Emergent Adverse Events (TEAEs)
Time Frame: Assessed starting from Day 1 of treatment to Day 113 in Dose Expansion phase.
Population: The Safety population comprised all randomised subjects who received any amount of study drug. Summaries, listings, and analyses were based on the treatment actually received. Screen failures and randomised subjects who did not receive any medication were excluded from the safety analysis set.
Measure: Count of Participants; unit: Participants
Groups:
- Dose Expansion EXN407 Cohort Study Eye; Dose Expansion EXN407 Cohort Contralateral Eye; Dose Expansion EXN407 Cohort Bilateral Eye: The highest well-tolerated dose of EXN407 will be evaluated where subjects will receive EXN407 at the selected dose or placebo twice a day for up to 84 days resulting in a total of 168 doses
  EXN407: EXN407 or placebo will be administered as a single 30 microliters drop twice a day, by unilateral eye drop administration to the study eye only.
- Dose Expansion Placebo Cohort Study Eye; Dose Expansion Placebo Cohort Contralateral Eye; Dose Expansion Placebo Cohort Bilateral Eye: Dose expansion cohort consisted of subjects randomised to receive EXN407 at the selected dose or placebo (vehicle) at a 2:1 drug: placebo ratio.
Arm/Group | Dose Expansion EXN407 Cohort Study Eye | Dose Expansion EXN407 Cohort Contralateral Eye | Dose Expansion EXN407 Cohort Bilateral Eye | Dose Expansion Placebo Cohort Study Eye | Dose Expansion Placebo Cohort Contralateral Eye | Dose Expansion Placebo Cohort Bilateral Eye
Number analyzed (Participants) | 23 | 23 | 23 | 12 | 12 | 12
Participants | 5 | 3 | 2 | 3 | 1 | 1

3. Secondary Outcome: To Evaluate the Systemic Pharmacokinetics of EXN407 Ophthalmic Solution in Subjects With DMO Secondary to Diabetes Mellitus by Tmax.
Description: Measured by characterizing the PK profile by estimating the time of the maximum plasma drug concentration (Tmax) of EXN407 in plasma.
Time Frame: Blood draws for PK will be collected only on Day 3(Dose Escalation) and Day 8(Dose Expansion) at the following timepoints: pre-dose and 15 mins, 30 mins, 1, 2, 3,and 4 hours post-dose.
Population: Number of participants with detectable values were analyzed. Limited quantifiable concentration-time data was available for this study, as such the plasma PK characteristics of EXN407, in particular the dose dependency, could not be comprehensively characterised. In the low dose group (0.5 mg/mL), PK parameters could not be determined due to a lack of quantifiable concentration-time data.
Measure: Mean (Standard Deviation); unit: hour
Groups:
- Dose Escalation: Cohort 1 (0.5 mg/mL) Day 3: Each subject will receive a low-dose 0.5 mg/mL (0.05%) of EXN407 or placebo twice a day in 14 doses over a 7 day period.
  EXN407: EXN407 or placebo will be administered as a single 30 microliters drop twice a day, by unilateral eye drop administration to the study eye only.
- Dose Escalation: Cohort 2 (1.0 mg/mL) Day 3: Each subject will receive a mid-dose 1 mg/mL (0.1%) of EXN407 or placebo twice a day in 14 doses over a 7 day period.
  EXN407: EXN407 or placebo will be administered as a single 30 microliters drop twice a day, by unilateral eye drop administration to the study eye only.
- Dose Escalation: Cohort 3 (1.5 mg/mL) Day 3: Each subject will receive a high-dose 1.5 mg/mL (0.15%) of EXN407 or placebo twice a day in 14 doses over a 7 day period.
  EXN407: EXN407 or placebo will be administered as a single 30 microliters drop twice a day, by unilateral eye drop administration to the study eye only.
- Dose Expansion Cohort (1.5 mg/mL) Day 8: The highest well-tolerated dose of EXN407 will be evaluated where subjects will receive EXN407 at the selected dose or placebo twice a day for up to 84 days resulting in a total of 168 doses
  EXN407: EXN407 or placebo will be administered as a single 30 microliters drop twice a day, by unilateral eye drop administration to the study eye only.
Arm/Group | Dose Escalation: Cohort 1 (0.5 mg/mL) Day 3 | Dose Escalation: Cohort 2 (1.0 mg/mL) Day 3 | Dose Escalation: Cohort 3 (1.5 mg/mL) Day 3 | Dose Expansion Cohort (1.5 mg/mL) Day 8
Number analyzed (Participants) | 2 | 3 | 3 | 22
hour | NA (NA) — Below the level of detection | 0.5 (0) | 0.5 (0.000000000123) | 0.494 (0.276)

4. Secondary Outcome: To Evaluate the Systemic Pharmacokinetics of EXN407 Ophthalmic Solution in Subjects With DMO Secondary to Diabetes Mellitus by Cmax
Description: Measured by characterizing the PK profile by estimating the maximum observed drug plasma concentration (Cmax) of EXN407 in plasma.
Time Frame: as for outcome 3
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Dose Escalation: Cohort 1 (0.5 mg/mL) Day 3 | Dose Escalation: Cohort 2 (1.0 mg/mL) Day 3 | Dose Escalation: Cohort 3 (1.5 mg/mL) Day 3 | Dose Expansion Cohort (1.5 mg/mL) Day 8
Number analyzed (Participants) | 2 | 3 | 3 | 22
ng/mL | NA (NA) — Below the level of detection | 0.0571 (0) | 0.0831 (0.0253) | 0.0883 (0.0410)

5. Secondary Outcome: To Evaluate the Systemic Pharmacokinetics of EXN407 Ophthalmic Solution in Subjects With DMO Secondary to Diabetes Mellitus by AUC.
Description: Measured by characterizing the PK profile by estimating the area under the curve (AUC) of EXN407 in plasma.
Time Frame: as for outcome 3
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: hr*ng/mL
Arm/Group | Dose Escalation: Cohort 1 (0.5 mg/mL) Day 3 | Dose Escalation: Cohort 2 (1.0 mg/mL) Day 3 | Dose Escalation: Cohort 3 (1.5 mg/mL) Day 3 | Dose Expansion Cohort (1.5 mg/mL) Day 8
Number analyzed (Participants) | 2 | 3 | 3 | 22
hr*ng/mL | NA (NA) — Below the level of detection | 0.0368 (0) | 0.153 (0.205) | 0.0845 (0.112)

6. Secondary Outcome: To Evaluate the Systemic Pharmacokinetics of EXN407 Ophthalmic Solution in Subjects With DMO Secondary to Diabetes Mellitus by t½.
Description: Measured by characterizing the PK profile by estimating the apparent elimination half-life (t½) of EXN407 in plasma.
Time Frame: as for outcome 3
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: hour
Arm/Group | Dose Escalation: Cohort 1 (0.5 mg/mL) Day 3 | Dose Escalation: Cohort 2 (1.0 mg/mL) Day 3 | Dose Escalation: Cohort 3 (1.5 mg/mL) Day 3 | Dose Expansion Cohort (1.5 mg/mL) Day 8
Number analyzed (Participants) | 2 | 3 | 3 | 22
hour | NA (NA) — Below the level of detection | 0 (0) | 0 (0) | 0 (0)

7. Secondary Outcome: To Evaluate Changes in Ocular Functional Measures as Assessed Using Ophthalmoscopy.
Description: Measured by the changes from baseline in ophthalmic examination finding through ophthalmoscopy (BCVA (Letters))
Time Frame: From Day 1 of Treatment to End of Treatment i.e. assessed upto 36 Days/EOS in Dose Escalation and upto 4 months(113 days/EOS) in Dose Expansion.
Measure: Mean (Standard Deviation); unit: BCVA (Letters)
Groups:
- Dose Escalation: Cohort 1 (0.5 mg/mL) Study Eye; Dose Escalation: Cohort 1 (0.5 mg/mL) Contralateral Eye: Each subject will receive a low-dose 0.5 mg/mL (0.05%) of EXN407 or placebo twice a day in 14 doses over a 7 day period.
  EXN407: EXN407 or placebo will be administered as a single 30 microliters drop twice a day, by unilateral eye drop administration to the study eye only.
- Dose Escalation: Cohort 2 (1.0 mg/mL) Study Eye; Dose Escalation: Cohort 2 (1.0 mg/mL) Contralateral Eye: Each subject will receive a mid-dose 1 mg/mL (0.1%) of EXN407 or placebo twice a day in 14 doses over a 7 day period.
  EXN407: EXN407 or placebo will be administered as a single 30 microliters drop twice a day, by unilateral eye drop administration to the study eye only.
- Dose Escalation: Cohort 3 (1.5 mg/mL) Study Eye; Dose Escalation: Cohort 3 (1.5 mg/mL) Contralateral Eye: Each subject will receive a high-dose 1.5 mg/mL (0.15%) of EXN407 or placebo twice a day in 14 doses over a 7 day period.
  EXN407: EXN407 or placebo will be administered as a single 30 microliters drop twice a day, by unilateral eye drop administration to the study eye only.
- Dose Expansion Cohort (1.5 mg/mL) Study Eye; Dose Expansion Cohort (1.5 mg/mL) Contralateral Eye: The highest well-tolerated dose of EXN407 will be evaluated where subjects will receive EXN407 at the selected dose or placebo twice a day for up to 84 days resulting in a total of 168 doses
  EXN407: EXN407 or placebo will be administered as a single 30 microliters drop twice a day, by unilateral eye drop administration to the study eye only.
Arm/Group | Dose Escalation: Cohort 1 (0.5 mg/mL) Study Eye | Dose Escalation: Cohort 1 (0.5 mg/mL) Contralateral Eye | Dose Escalation: Cohort 2 (1.0 mg/mL) Study Eye | Dose Escalation: Cohort 2 (1.0 mg/mL) Contralateral Eye | Dose Escalation: Cohort 3 (1.5 mg/mL) Study Eye | Dose Escalation: Cohort 3 (1.5 mg/mL) Contralateral Eye | Pooled Placebo (Cohort 1, Cohort 2, Cohort 3) Study Eye | Pooled Placebo (Cohort 1, Cohort 2, Cohort 3) Contralateral Eye | Dose Expansion Cohort (1.5 mg/mL) Study Eye | Dose Expansion Cohort (1.5 mg/mL) Contralateral Eye | Dose Expansion Placebo Cohort Study Eye | Dose Expansion Placebo Cohort Contralateral Eye
Number analyzed (Participants) | 3 | 3 | 3 | 3 | 3 | 3 | 4 | 4 | 23 | 23 | 12 | 12
BCVA (Letters) | -5.0 (8.72) | -5.0 (9.54) | -2.0 (2.65) | -1.0 (3.61) | 3.0 (2.0) | -4.0 (7.94) | -1.3 (3.3) | -3.0 (5.35) | -0.1 (3.54) | -1.7 (6.06) | 1.3 (5.14) | 1.3 (5.31)

8. Secondary Outcome: To Evaluate Changes in Ocular Structural Measures as Assessed Using Ophthalmoscopy.
Description: Measured by the changes from baseline in ophthalmic examination finding through ophthalmoscopy (corneal thickness).
Time Frame: From Day 1 of Treatment to End of Treatment i.e. assessed upto 36 Days/EOS in Dose Escalation and up to 4 months(113 days) in Dose Expansion.
Measure: Mean (Standard Deviation); unit: corneal thickness (microns)
Arm/Group | Dose Escalation: Cohort 1 (0.5 mg/mL) Study Eye | Dose Escalation: Cohort 1 (0.5 mg/mL) Contralateral Eye | Dose Escalation: Cohort 2 (1.0 mg/mL) Study Eye | Dose Escalation: Cohort 2 (1.0 mg/mL) Contralateral Eye | Dose Escalation: Cohort 3 (1.5 mg/mL) Study Eye | Dose Escalation: Cohort 3 (1.5 mg/mL) Contralateral Eye | Pooled Placebo (Cohort 1, Cohort 2, Cohort 3) Study Eye | Pooled Placebo (Cohort 1, Cohort 2, Cohort 3) Contralateral Eye | Dose Expansion Cohort (1.5 mg/mL) Study Eye | Dose Expansion Cohort (1.5 mg/mL) Contralateral Eye | Dose Expansion Placebo Cohort Study Eye | Dose Expansion Placebo Cohort Contralateral Eye
Number analyzed (Participants) | 3 | 3 | 3 | 3 | 3 | 3 | 4 | 4 | 23 | 23 | 12 | 12
corneal thickness (microns) | -5.0 (6.93) | -2.7 (8.33) | 15.3 (7.02) | 11.0 (19.08) | -3.0 (4.00) | -10.3 (18.93) | -0.8 (3.77) | 1.3 (4.50) | 0.2 (8.61) | 0.1 (10.52) | 2.4 (11.27) | 0.5 (11.35)

ADVERSE EVENTS:
Time Frame: Each subject in the Dose Escalation cohorts (numbered Cohorts 1, 2, 3, etc.) received EXN407 or vehicle BID over a 7-day period Each subject in the Dose Expansion received EXN407 or vehicle BID over an 84-day period
Description: Assessed starting from Day 1 of treatment to Day 36 in Dose Expansion phase. Assessed starting from Day 1 of treatment to Day 113 in Dose Expansion phase. Arms/Groups are combined (not separated into study eye and fellow eye) as both ocular and non-ocular adverse events are reported.
Arm/Group | Dose Escalation EXN407 Cohort 1 | Dose Escalation EXN407 Cohort 2 | Dose Escalation EXN407 Cohort 3 | Dose Escalation Pooled Placebo Cohort | Dose Expansion EXN407 Cohort | Dose Expansion Placebo Cohort
All-Cause Mortality (participants affected / at risk) | 0/3 | 0/3 | 0/3 | 0/4 | 0/23 | 0/12
Serious Adverse Events (participants affected / at risk) | 0/3 | 0/3 | 0/3 | 0/4 | 2/23 | 1/12
Other Adverse Events (participants affected / at risk) | 2/3 | 2/3 | 1/3 | 1/4 | 11/23 | 9/12
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dose Escalation EXN407 Cohort 1 (N=3) | Dose Escalation EXN407 Cohort 2 (N=3) | Dose Escalation EXN407 Cohort 3 (N=3) | Dose Escalation Pooled Placebo Cohort (N=4) | Dose Expansion EXN407 Cohort (N=23) | Dose Expansion Placebo Cohort (N=12)
Angina pectoris (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) — single instance of moderate angina pectoris (atypical chest pain) that was assessed as unlikely related to the study drug. The study drug was interrupted, and the event resolved within 23 days
non-ST elevation acute coronary syndrome (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) — single instance of severe acute coronary syndrome (non-ST elevation acute coronary syndrome) that was assessed as unlikely related to the study drug. The study drug was interrupted, and the event resolved within 10 days.
severe hypoglycaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) — single instance of severe hypoglycaemia (severe hypoglycaemia) that was assessed as unlikely related to the study drug. The study drug was not changed, and the event resolved within 1 day without treatment.
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | Dose Escalation EXN407 Cohort 1 (N=3) | Dose Escalation EXN407 Cohort 2 (N=3) | Dose Escalation EXN407 Cohort 3 (N=3) | Dose Escalation Pooled Placebo Cohort (N=4) | Dose Expansion EXN407 Cohort (N=23) | Dose Expansion Placebo Cohort (N=12)
Blepharitis (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) — 1 subject in the 0.5 mg/mL EXN407 cohort (#108-001) had 1 event of mild seborrheic blepharitis (bilateral affecting both eyes)
Posterior capsule opacification (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) — 1 subject in the 1.0 mg/mL group (#109-004) had 1 event of right posterior capsule opacification (bilateral affecting both eyes).
Vision blurred (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) — 1 subject in the 0.5 mg/mL EXN407 cohort (#106-006) had 1 event of blurred vision in mornings (bilateral affecting both eyes).
Eye pruritus (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) — 2 subjects in the EXN407 group (#103-009 and #108-018) had 2 events (1 event each in study eye) of eye pruritis (left itchy eye and right itchy eye, respectively).
Hypoglycemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 1 (1) | 0/2 (0) | 0 (0) | 1 (1)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
COVID-19 (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0)
C-reactive protein increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Episcleritis (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) — Episcleritis. 1 subject in the placebo group (#112-006) had 1 event of episcleritis right eye (study eye).
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) — Dizziness
Lower respiratory tract infection (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Gastrointestinal infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Nasopharyngitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Otitis media (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Visual field defect (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Migraine (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Blood phosphorus decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Electrocardiogram ST segment elevation (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Punctate keratiis (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) — 1 subject in the placebo group (#108-024) had 1 event of punctate epithelial erosions right eye (study eye).
Foreign body sensation in eyes (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) — 1 subject in the placebo group (#112-002) had 1 event of foreign body sensation right eye (study eye).
Cataract cortical (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) — 1 subject in the placebo group (#108-015) had 1 event of increase in degree of cortical cataract (bilateral affecting both eyes).
Eye irritation (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) — 1 subject in the placebo group (#112-002) had 1 event of irritation - right eye (study eye).
Hyperglycemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Sinus bradycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Lymphadenopathy (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Acrochordon (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-01-28): https://cdn.clinicaltrials.gov/large-docs/56/NCT04565756/Prot_SAP_000.pdf